CLINICAL TRIAL: NCT06721494
Title: A Phase 2 Single-Dose Study to Evaluate Safety and Efficacy of CS-1103 in Participants With Methamphetamine Use Disorder Not Seeking Treatment Receiving a Single Dose of Methamphetamine
Brief Title: A Single-Dose Study to Evaluate Safety and Efficacy of CS-1103 in Participants Receiving a Single Dose of Methamphetamine
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Clear Scientific, Inc. (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CS-1103-02; 5U01DA058548-02 (NIH)
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Methamphetamine Intoxication; Methamphetamine Disorders; Methamphetamine Abuse
MeSH Terms: interventions — Methamphetamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants receive methamphetamine HCl (30 mg) followed by placebo (saline).
  Interventions: Drug: Methamphetamine; Drug: Sterile Saline
- Active (Active Comparator): Participants receive methamphetamine HCl (30 mg) followed by one of four doses of CS-1103
  Interventions: Drug: Methamphetamine; Drug: CS-1103

INTERVENTIONS:
Drug: Methamphetamine — Methamphetamine HCl for intravenous administration
Drug: Sterile Saline — Sterile Saline for intravenous administration
  Arms: Placebo
Drug: CS-1103 — CS-1103 for intravenous administration
  Arms: Active

SUMMARY:
The purpose of the study is to evaluate the safety, efficacy, and pharmacokinetics of four single, increasing doses of CS-1103, given by intravenous (IV) infusion in otherwise healthy, non-treatment seeking participants with methamphetamine use disorder in the presence of a clinically relevant dose of methamphetamine HCl (30 mg IV).

ELIGIBILITY:
Major Inclusion Criteria:

1. Healthy participants aged 18 to 55 years, inclusive;
2. Meets DSM-5 criteria for methamphetamine use disorder;
3. Not seeking treatment for methamphetamine use disorder;
4. Primary route of methamphetamine self-administration must be intravenous or smoking;
5. Able to abstain from methamphetamine without experiencing severe withdrawal;
6. A body mass index between 18 to 30 kg/m2, inclusive and a minimum body weight of 50 kg;
7. Females must not be lactating and must have a negative pregnancy test during screening and admission.

Major Exclusion Criteria:

1. Estimated glomerular filtration rate <60 mL/min/1.73 m2;
2. History of cardiovascular disease;
3. Current moderate to severe use disorder for alcohol, cannabis, cocaine, opioids, or benzodiazepines;
4. History of any clinically important disease or disorder which, in the opinion of the Investigator, may interfere with safe study participation.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-02-05 (Estimated); Primary Completion 2026-09-04 (Estimated); Study Completion 2026-09-11 (Estimated)

PRIMARY OUTCOMES:
Number of participants with CS-1103-related adverse events (AEs) assessed by physical examinations | 3 days plus follow-up on Day 10
  Physical examinations
Number of participants with CS-1103-related adverse events (AEs) assessed by electrocardiograms (ECGs) | 3 days plus follow-up on Day 10
  Digital 12-lead electrocardiograms (ECGs). Any correlation between CS-1103 plasma concentrations and changes in QT intervals will be noted.
Number of participants with CS-1103-related adverse events (AEs) assessed by vital signs | 3 days plus follow-up on Day 10
  Blood pressure, pulse rate, respiratory rate, oxygen saturation, and body temperature
Number of participants with CS-1103-related adverse events (AEs) assessed by laboratory parameters | 3 days plus follow-up on Day 10
  Clinical chemistry, hematology, coagulation, and urinalysis
Time course and magnitude of urine excretion of methamphetamine | 48 hours
  Measurement of concentration of methamphetamine in urine

SECONDARY OUTCOMES:
Time course of CS-1103 blood and urine concentrations | 48 hours
  Measurement of plasma and urine concentrations of CS-1103

CONTACTS AND LOCATIONS:
Overall Officials: Xinhua Li, Ph.D., Principal Investigator — Clear Scientific, Inc.
Locations (1):
- California Clinical Trials Medical Group, Glendale, California, United States